CLINICAL TRIAL: NCT02021409
Title: A Randomized, Parallel Group, Open-label, Multicenter Study to Investigate the Efficacy and Safety of Oral BAY85-3934 and Active Comparator (Darbepoetin Alfa) in the Maintenance Treatment of Anemia in Pre-dialysis Subjects With Chronic Kidney Disease on Darbepoetin Treatment in Europe and Asia Pacific
Brief Title: Maintenance Treatment of Anemia in Pre-dialysis Subjects With Chronic Kidney Disease on Darbepoetin Treatment Versus BAY85-3934
Acronym: DIALOGUE 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15261; 2013-001192-21 (EudraCT Number)
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Anemia; Renal Insufficiency, Chronic
Keywords: Anemia on CKD
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BAY85-3934 (25mg) (Experimental): Fixed starting dose of 25 mg of BAY85-3934 oral tablet (once daily dose) titrated at the scheduled dose control visits. Titration occuring every 4-weeks will be based on the subject's hemoglobin (Hb) response and tolerability of the prior dose. Total treatment time is 16 weeks. Planned doses include 15, 25, 50, 75, 100, and 150 mg once daily.
  Interventions: Drug: BAY85-3934
- BAY85-3934 (50mg) (Experimental): Fixed starting dose of 50 mg of BAY85-3934 oral tablet (once daily dose) titrated at the scheduled dose control visits. Titration occuring every 4-weeks will be based on the subject's Hb response and tolerability of the prior dose. Total treatment time is 16 weeks. Planned doses include 15, 25, 50, 75, 100, and 150 mg once daily.
  Interventions: Drug: BAY85-3934
- BAY85-3934 (75mg) (Experimental): Fixed starting doses of 75 mg of BAY85-3934 oral tablet (once daily dose) titrated at the scheduled dose control visits. Titration occuring every 4-weeks will be based on the subject's Hb response and tolerability of the prior dose. Total treatment time is 16 weeks. Planned doses include 15, 25, 50, 75, 100, and 150 mg once daily.
  Interventions: Drug: BAY85-3934
- Darbepoetin alfa (Active Comparator): Darbepoetin (intravenous or subcutaneous) will be administered according to the local label and titrated at the scheduled dose control visits. Titration will be based on the subject's Hb response and tolerability of the prior dose.
  Interventions: Biological: Darbepoetin alfa

INTERVENTIONS:
Drug: BAY85-3934 — Oral doses of BAY 85-3934 will be available in multiples of 5, 25, and 75 mg tablets
  Arms: BAY85-3934 (25mg); BAY85-3934 (50mg); BAY85-3934 (75mg)
Biological: Darbepoetin alfa
  Arms: Darbepoetin alfa

SUMMARY:
Anaemia is a condition in which blood has a lower than normal number of red blood cells. It can also occur if red blood cells do not contain enough haemoglobin, an oxygen carrying part of blood. Anaemia is common in patients with chronic kidney disease. Healthy kidneys produce a hormone called erythropoietin, which stimulates the bone marrow to produce the proper number of red blood cells needed to carry oxygen to vital organs. Chronic kidney disease is a general term that means that the kidneys are not functioning to their full potential. The study drug, BAY85-3934, is being evaluated as a drug to increase the body's ability to produce erythropoietin.

The purpose of this study is to find out if the study drug, a tablet taken orally, is safe and effective for the treatment of anaemia associated with chronic kidney disease.

The study will enroll 120 patients at multiple locations in Europe, Asia and Australia. Participation will involve a screening visit and between 12 and 15 study visits scheduled over a period of approximately 5 to 7 months. The estimated total duration of study treatment will be 16 weeks. During these scheduled visits patients will undergo a number of procedures to confirm efficacy and safety of the study drug, including measurement of heart rate and blood pressure, physical examination, Electrocardiogram and blood/urine sample collection for laboratory tests.

The study will be conducted at 3 hospitals in the UK. Bayer HealthCare AG is funding this research.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age with anemia of chronic kidney disease (CKD) at screening
* Estimated glomerular filtration rate (eGFR) of < 60 mL/min/1.73 m2 (Modification of Diet in Renal Disease or the formula according to Matsuo, et al.)
* Not on dialysis and not expected to begin dialysis during the treatment period of the study (at least 16 weeks from randomization)
* Treated with darbepoetin via intravenous (IV) or subcutaneous (SC) route with a weekly, bi-weekly, or monthly dose, having had no more than one dose change within 8 weeks prior to randomization
* At least one kidney
* Mean screening hemoglobin (Hb) concentration of 10.0 to 12.0 g/dL
* Men who agree to use adequate contraception when sexually active or women without childbearing potential

Exclusion Criteria:

* Subjects with significant acute or chronic bleeding, such as overt gastrointestinal bleeding
* Active hemolysis or diagnosis of hemolytic syndrome
* History of myelodysplastic syndrome, multiple myeloma, marrow fibrosis, or pure red-cell aplasia (PRCA)
* History of hemosiderosis or hemochromatosis
* Hereditary hemoglobinopathies (such as sickle cell disease and thalassemia major)
* Aplastic anemia
* Chronic lymphoproliferative diseases
* Proliferative choroidal or retinal disease, such as neovascular age-related macular degeneration or proliferative diabetic retinopathy that is likely to require invasive treatment (intraocular injections or laser photocoagulation) during the study
* Chronic inflammatory disease that could impact erythropoiesis (e.g., systemic lupus erythematosis, rheumatoid arthritis, celiac disease) even if it is currently in remission
* Known hypersensitivity to the study drugs (active substances or excipients of the preparations)
* Uncontrolled and symptomatic hyperparathyroidism
* Uncontrolled active infection
* Previous or concurrent cancer except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis, and T1) or any cancer curatively treated > 3 years prior to randomization
* Any allograft (including renal allograft) in place and on immunosuppressive therapy or a scheduled kidney transplant within the next 16 weeks (being on a waiting list does not exclude the subject)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2015-10-15 (Actual); Study Completion 2015-11-23 (Actual)

PRIMARY OUTCOMES:
Change in local laboratory hemoglobin level from baseline to the average during the last 4 weeks treatment period | Baseline and week 12 to 16

SECONDARY OUTCOMES:
Maintenance in hemoglobin target range (10.0 to 12.0 g/dL) | Up to 16 weeks
Change in hemoglobin level | Baseline up to 16 weeks
Number of patients with hemoglobin levels outside the target range | Week 12 to 16
Dose level in the evaluation period | Week 12 to 16
Duration of exposure on each dose level | Up to 16 weeks
Number of subjects requiring titration of dose | Up to 16 weeks
Number of participants with serious adverse events as a measure of safety and tolerability | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (50):
- Australia (2):
  - Gosford, New South Wales
  - Reservoir, Victoria
- Bulgaria (6):
  - Dobrich
  - Lovech
  - Montana
  - Pazardzhik
  - Sofia
  - Stara Zagora
- France (2):
  - Grenoble
  - Pierre-Bénite
- Bonn, North Rhine-Westphalia, Germany
- Hungary (6):
  - Baja
  - Budapest
  - Esztergom
  - Kaposvár
  - Pécs
  - Szigetvár
- Israel (4):
  - Ashkelon
  - Hadera
  - Kfar Saba
  - Nahariya
- Italy (6):
  - Napoli, Campania
  - Brescia, Lombardy
  - Cremona, Lombardy
  - Lecco, Lombardy
  - Pavia, Lombardy
  - Livorno, Tuscany
- Japan (9):
  - Kitakyushu, Fukuoka
  - Ōkawa, Fukuoka
  - Muroran, Hokkaido
  - Morioka, Iwate
  - Fujisawa, Kanagawa
  - Kuwana, Mie-ken
  - Chiba
  - Fukuoka
  - Nagano
- Poland (2):
  - Bialystok
  - Radom
- Romania (3):
  - Bucharest
  - Oradea
  - Târgu Mureş
- Bucheon-si, Gyeonggido, South Korea
- Spain (3):
  - L'Hospitalet de Llobregat, Barcelona
  - San Sebastián de los Reyes, Madrid
  - Madrid
- Turkey (Türkiye) (3):
  - Ankara Univ. Medical Faculty, Ankara
  - Baskent University Medical Faculty, Ankara
  - Sifa University Medical Faculty, Izmir
- United Kingdom (2):
  - Cambridge, Cambridgeshire
  - Liverpool

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- See also: Click here and search for results provided by EudraCT — https://www.clinicaltrialsregister.eu/
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/